CLINICAL TRIAL: NCT00107497
Title: Prospective Randomised Clinical Trial Testing 5.7 Gy and 6.0 Gy Fractions of Whole Breast Radiotherapy in Terms of Late Normal Tissue Responses and Tumour Control - FAST
Brief Title: Radiation Therapy in Treating Women With Localized Breast Cancer
Acronym: FAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000417730; ICR-04/MRE06/17 (Other Grant/Funding Number: UK MREC)
Record Dates: First submitted 2005-04-05; First posted 2005-04-06 (Estimated); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Active Comparator): 50Gy in 25 fractions of radiation therapy over 5 weeks
  Interventions: Radiation: Radiation therapy
- Test group 1 (Active Comparator): 30Gy in 5 fractions of radiation therapy over 5 weeks
  Interventions: Radiation: Radiation therapy
- Test group 2 (Active Comparator): 28.5Gy in 5 fractions of radiation therapy over 5 weeks
  Interventions: Radiation: Radiation therapy

INTERVENTIONS:
Radiation: Radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill tumor cells. Giving radiation therapy in different ways and giving it after surgery may kill any tumor cells that remain after surgery.

PURPOSE: This randomized clinical trial is studying radiation therapy to see how well it works in treating women with localized breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare late normal tissue effects of standard vs 2 different dose levels of hypofractionated adjuvant whole breast radiotherapy, in terms of changes in photographic breast appearance, in women with localized breast cancer who are at average or low risk of recurrence.
* Compare tumor control in patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to participating center. Patients are randomized to 1 of 3 treatment arms.

* Arm I (control): Patients undergo standard radiotherapy 5 days a week for 5 weeks.
* Arm II: Patients undergo hypofractional radiotherapy once a week for 5 weeks.
* Arm III: Patients undergo hypofractional radiotherapy (at a lower dose than arm II) once a week for 5 weeks.

After completion of study treatment, patients are followed annually for 5-10 years.

PROJECTED ACCRUAL: A total of 900 patients (300 per treatment arm) will be accrued for this study within 12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of invasive carcinoma of the breast

  * Localized disease

    * Pathological tumor size < 3.0 cm in diameter
    * Axillary node negative
* At average or low risk of local tumor recurrence
* Must have undergone prior breast-preserving surgery

  * No prior mastectomy
  * Complete microscopic resection of tumor
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* 50 and over

Sex

* Female

Menopausal status

* Not specified

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior neoadjuvant or adjuvant cytotoxic chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* No concurrent lymphatic radiotherapy
* No concurrent radiotherapy boost to the breast

Surgery

* See Disease Characteristics

Ages: 50 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 917 (Actual)
Dates: Start 2004-10-05 (Actual); Primary Completion 2007-03-09 (Actual); Study Completion 2017-03-09 (Actual)

PRIMARY OUTCOMES:
Change in photographic breast appearance | 2 years post randomisation
  Change in photographic breast appearance at 2 years post randomisation compared to a baseline pre-surgical photograph

CONTACTS AND LOCATIONS:
Overall Officials: John R. Yarnold, MD, FRCR, Study Chair — Royal Marsden NHS Foundation Trust
Locations (19):
- United Kingdom (19):
  - Sussex Cancer Centre at Royal Sussex County Hospital, Brighton, England
  - Cumberland Infirmary, Carlisle, England
  - Cheltenham General Hospital, Cheltenham, England
  - Royal Devon and Exeter Hospital, Exeter, England
  - Ipswich Hospital NHS Trust, Ipswich, England
  - Christie Hospital NHS Trust, Manchester, England
  - Clatterbridge Centre for Oncology NHS Trust, Merseyside, England
  - Berkshire Cancer Centre at Royal Berkshire Hospital, Reading, England
  - Royal Shrewsbury Hospital, Shrewsbury, England
  - University Hospital of North Staffordshire, Stoke-on-Trent, England
  - Royal Marsden NHS Foundation Trust - Surrey, Sutton, England
  - Torbay Hospital, Torquay Devon, England
  - Royal Cornwall Hospital, Truro, Cornwall, England
  - Southend University Hospital NHS Foundation Trust, Westcliff-on-Sea, England
  - Worcester Royal Hospital, Worcester, England
  - Worthing Hospital, Worthing, England
  - Velindre Cancer Center at Velindre Hospital, Cardiff, Wales
  - Halton Hospital - North Cheshire Hospitals NHS Trust, Cheshire
  - Hereford Hospitals NHS Trust, Hereford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brunt AM, Haviland JS, Sydenham M, Agrawal RK, Algurafi H, Alhasso A, Barrett-Lee P, Bliss P, Bloomfield D, Bowen J, Donovan E, Goodman A, Harnett A, Hogg M, Kumar S, Passant H, Quigley M, Sherwin L, Stewart A, Syndikus I, Tremlett J, Tsang Y, Venables K, Wheatley D, Bliss JM, Yarnold JR. Ten-Year Results of FAST: A Randomized Controlled Trial of 5-Fraction Whole-Breast Radiotherapy for Early Breast Cancer. J Clin Oncol. 2020 Oct 1;38(28):3261-3272. doi: 10.1200/JCO.19.02750. Epub 2020 Jul 14. PMID 32663119
- See also: First results of the randomised UK FAST Trial of radiotherapy hypofractionation for treatment of early breast cancer (CRUKE/04/015), Radiotherapy and Oncology, Volume 100, Issue 1, 2011, Pages 93 - 100 — https://doi.org/10.1016/j.radonc.2011.06.026